CLINICAL TRIAL: NCT06180109
Title: An Open-label, Balanced, Randomized, Two Treatment, Two Sequence, Two Period, Two Way Cross-over, Single Oral Dose Bioequivalence Study of Empagliflozin 25 mg Film Coated Tablets of Humanis, Turkey and Jardiance (Empagliflozin) 25 mg Film-coated Tablets of Boehringer Ingelheim International GmbH, Germany in Normal, Healthy, Adult, Human Subjects Under Fasting Condition
Brief Title: Bioequivalence Study of Empagliflozin 25 mg Film Coated Tablets of Humanis, Turkey and Jardiance (Empagliflozin) 25 mg Film-coated Tablets of Boehringer Ingelheim International GmbH, Germany in Normal, Healthy, Adult, Human Subjects Under Fasting Condition
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Humanis Saglık Anonim Sirketi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: PR/BE/22/266
Record Dates: First submitted 2023-12-06; First posted 2023-12-22 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Type2 Diabetes Mellitus
MeSH Terms: interventions — empagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Empagliflozin film coated tablets (Experimental): Empagliflozin 25 mg film coated tablets
  Interventions: Drug: Empagliflozin film coated tablets; Drug: Jardiance film-coated tablets
- Jardiance film-coated tablets (Active Comparator): Jardiance (Empagliflozin) 25 mg film-coated tablets
  Interventions: Drug: Empagliflozin film coated tablets; Drug: Jardiance film-coated tablets

INTERVENTIONS:
Drug: Empagliflozin film coated tablets — 1 film coated tablet of 25 mg Empagliflozin
Drug: Jardiance film-coated tablets — 1 film coated tablet of 25 mg Empagliflozin

SUMMARY:
An open-label, balanced, randomized, two treatment, two sequence, two period, two way cross-over, single oral dose bioequivalence study of Empagliflozin 25 mg film coated tablets of Humanis, Turkey and Jardiance (Empagliflozin) 25 mg film-coated tablets of Boehringer Ingelheim International GmbH, Germany in normal, healthy, adult, human subjects under fasting condition.

ELIGIBILITY:
Inclusion Criteria:

Willing to provide written informed consent for participation in the study, and an ability to comprehend the nature and purpose of the study;

* Willing to be available for the entire study period and to comply protocol requirements;
* Normal, healthy, adult, human subject of 18-45 years (both inclusive) of age;
* Body mass index in the range of 18.50 - 30.00 kg/m2 (both inclusive);
* Normal health status as determined by baseline medical and medication history, at the time of screening and vital signs measurements and physical examination at the time of screening as well as check-in of each study period;
* Normal or clinically non-significant laboratory values as determined by hematological, biochemistry tests and urine analysis;
* Normal or clinically non-significant 12-lead ECG recording;
* Non-smokers and willing to abstain from chewing any tobacco containing products at least 72.00 hours prior to check-in until last sample collection in each study period;
* Non Alcoholic;
* Willing to abstain from xanthine or its derivative containing food or beverages (e.g. chocolates, tea, coffee or cola drinks), at least 48.00 hours prior to check-in until last sample collection in each study period;
* Willing to abstain from grapefruit or its juice at least 72.00 hours prior to check-in until last sample collection in each study period;
* For female subjects:
* Negative urine pregnancy test during screening and negative serum β-hCG test at the time of check-in of each study period;
* Female subjects with child bearing potential or those within their first two years of onset of menopausal syndrome willing to either abstain from sexual intercourse, or should use of acceptable birth control methods for at least 15 days before 1st check-in till 15 days post last-dose / entire study period. [Acceptable birth control methods include barrier methods such as diaphragm/condom with or without spermicide or surgically sterile (bilateral tubal ligation, bilateral oophorectomy or hysterectomy has been performed)].

Exclusion Criteria:

Any medical or surgical conditions, which might significantly interfere with the functioning of gastrointestinal tract and of blood forming organs;

* Significant history or current evidence of malignancy or chronic - infectious, cardiovascular, renal, hepatic, ophthalmic, pulmonary, neurological, metabolic (endocrine), hematological, gastrointestinal, dermatological, immunological or psychiatric diseases, or organ dysfunction;
* History of diabetes mellitus or insulin resistance.
* Any major illness or hospitalized within 90 days prior to the first check-in;
* Requiring medication for any ailment having enzyme-modifying activity within one month prior to first check-in and throughout the study;
* Use of any depot injection or an implant of any drug within 3 months prior to first check-in and throughout the study;
* Use of any prescribed medication (including herbal medicines and vitamin supplements) or OTC products within 30 days prior to first check-in and throughout the study;
* History or presence of significant gastric and/or duodenal ulceration;
* Difficulty in swallowing tablets or capsules;
* Use of any recreational drug or history of drug addiction;
* Participated in any clinical investigation requiring repeated blood sampling or have donated blood in past 90 days prior to first check-in;
* Positive urine alcohol and/or urine drug of abuse tests during check-in of each study period;
* Reactive test for Human Immunodeficiency Virus (HIV) type I/II antibodies or Hepatitis B surface antigen (HBsAg) or Hepatitis C virus antibodies;
* Lactating or nursing female subjects;
* Female subjects using hormonal contraceptive (either oral/implants);
* History of allergy or hypersensitivity intolerance to Empagliflozin or its formulation excipients which, in the opinion of a clinical investigator, would compromise the safety of the subject or the study;
* History of difficulty in accessibility of veins in arms.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2023-07-30 (Actual); Primary Completion 2023-08-27 (Actual); Study Completion 2023-10-06 (Actual)

PRIMARY OUTCOMES:
Maximum concentration obtained (Cmax) | 48 hours
  Two-sided 90% confidence intervals for ratio (test/reference) of the population means is within 80.00% to 125.00% for each of the Ln-transformed data Cmax
AUC from the 0 to infinity (AUC0-inf) | 48 hours
  Descriptive Statistics
Time of the maximum measured plasma concentration (Tmax) | 48 hours
  Descriptive Statistics

CONTACTS AND LOCATIONS:
Overall Officials: Hakan Gürpınar, Study Director — Humanis Saglık
Locations (1):
- Raptim Research Pvt. Ltd.,, Navi Mumbai, India

IPD SHARING:
Plan to Share IPD: No